CLINICAL TRIAL: NCT00361218
Title: Serum Brain-Derived Neurotrophic Factor (BDNF) and QEEG as Biological Markers of Response to (Es)Citalopram Treatment in Major Depressive Disorder
Brief Title: Biological Markers of Response to Treatment in Major Depressive Disorder
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Responsible Party: Principal Investigator, John W. Denninger, MD, PhD, Instructor in Psychiatry, Massachusetts General Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2005P000413
Record Dates: First submitted 2006-08-04; First posted 2006-08-08 (Estimated); Results first posted 2013-09-26 (Estimated); Last update posted 2018-05-11 (Actual); Status verified 2018-04

CONDITIONS: Major Depressive Disorder
Keywords: depression; biology
MeSH Terms: conditions — Depressive Disorder, Major; Depression | interventions — Escitalopram; Citalopram

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- open-label selective serotonin reuptake inhibitor (SSRI) (Other): citalopram or escitalopram
  Interventions: Drug: open-label selective serotonin reuptake inhibitor (SSRI)

INTERVENTIONS:
Drug: open-label selective serotonin reuptake inhibitor (SSRI) — Duration is 8 weeks. For escitalopram, starting dose is 10mg po qd,which can be increased up to 30mg po qd per clinical discretion. For citalopram, starting dose is 20mg po qd, which can be increased up to 60mg po qd per clinical discretion.
  Other Names: escitalopram or citalopram

SUMMARY:
The purpose of this study is to find out if two tests are useful in predicting whether someone with depression will get better when he or she is treated with an FDA approved antidepressant medication (either citalopram or escitalopram).

DETAILED DESCRIPTION:
Major depressive disorder (MDD) is a severe form of depression. MDD can significantly interfere with an individual's thoughts, behavior, mood, and physical health. People who suffer from MDD often experience feelings of worthlessness; they may feel hopeless and may be unable to cope with problems in their life. In addition, they often experience sleep disruption, loss of appetite, and chronic pain.

It often takes several weeks to find out if an antidepressant medication is going to work for someone. This research study aims to identify tests that are able to predict if a medication will work, even before a person starts to feel better. The first test is a measurement of the blood protein Brain-Derived Neurotrophic Factor (BDNF), which is involved with brain cell growth. The second test is a Quantitative Electroencephalogram (QEEG), which measures brain activity.

The study lasts for 8 weeks and involves 5 total visits to the clinic. Throughout the study, all subjects will receive either escitalopram (Lexapro) or citalopram (Celexa) on the basis of the study doctor's clinical judgment. The dose of the medications can be increased at any point in time if the study doctor thinks it is appropriate. After the first screen visit (which lasts about 3 hours), each subsequent half-hour visit will involve a 2-tablespoon blood draw to measure BDNF levels, as well as a QEEG in which small, painless electrodes are stuck to the subject's forehead and electrical activity of the brain is measured. At the end of the 8 weeks, subjects are offered 3 months of free follow-up care, including medications.

ELIGIBILITY:
Inclusion Criteria:

* Ages 18-65
* Meet criteria for current Major Depressive Disorder
* Antidepressant medication-free for at least 2 weeks prior to the start of the study

Exclusion Criteria:

* Pregnant or breastfeeding women
* Anyone who is suicidal
* Anyone with an unstable medical condition (cardiovascular, hepatic, renal, respiratory, endocrine, neurological, or hematological), substance abuse problem within the past 6 months, psychoses (past or current), hypothyroidism, or hypomania
* Anyone currently taking an SSRI
* Past intolerance to Lexapro or Celexa

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 72 (Actual)
Dates: Start 2005-10; Primary Completion 2008-12 (Actual); Study Completion 2008-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: John Denninger, MD, PhD, Principal Investigator — Depression Clinical and Research Program, Massachusetts General Hospital

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subjects were recruited from Boston/Salem Metropolitan Area via advertising on newspapers, television and radio, referrals from other clinicians, and patients who came into the Depression Research Program to participate in other studies
Pre-assignment Details: After consenting to participate, subjects were screened for the study and, if found to be eligible, returned for their baseline visit after one week, during which no psychotropic medication was allowed.
Period: Overall Study
Arm/Group | Open-label Selective Serotonin Reuptake Inhibitor (SSRI)
Started | 53 (met eligibility criteria and enrolled in the study)
Completed Baseline Assessment | 47
Completed | 30
Not Completed | 23
Not completed — Lost to Follow-up | 11
Not completed — Personal Reasons | 7
Not completed — terminated / withdrawn due to toxicity / | 5

BASELINE CHARACTERISTICS:
Groups:
- Open-label SSRI: citalopram or escitalopram
  open-label SSRI : Duration is 8 weeks. For escitalopram, starting dose is 10mg po qd,which can be increased up to 30mg po qd per clinical discretion. For citalopram, starting dose is 20mg po qd, which can be increased up to 60mg po qd per clinical discretion.
Arm/Group | Open-label SSRI
Number analyzed (Participants) | 47
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 46
  >=65 years | 1
Age, Continuous [Mean (Standard Deviation); unit: years] | 43.3 (13.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 25
  Male | 22
Region of Enrollment [Number; unit: participants]
  United States | 47

OUTCOME MEASURES:

1. Primary Outcome: Serum Brain-derived Neurotrophic Factor (BDNF) Levels
Description: "Pre-SSRI BDNF Level" refers to the data collection point before SSRI intake and "Post-SSRI BDNF Level" refers to the data collection point 8 weeks after SSRI intake.
Time Frame: 8 weeks
Measure: Mean (Standard Deviation); unit: pg/mL
Arm/Group | Open-label Selective Serotonin Reuptake Inhibitor (SSRI)
Number analyzed (Participants) | 28
pg/mL
  Pre-SSRI BDNF Level | 6077.270 (4371.67)
  Post-SSRI BDNF Level | 4393.24 (3263.70)

2. Primary Outcome: Quantitative Electroencephalogram (QEEG) Parameters as Predictors of Response
Description: Pre-treatment quantitative electroencephalogram (QEEG) refers to the data collection point before selective serotonin reuptake inhibitor (SSRI) treatment and Post-treatment QEEG refers to the data collection point 8 weeks after SSRI treatment initiation.
  Response refers to a greater than 50% decrease in Hamiton Depression Rating Scale from baseline, which ranges from 0 (no depression) to a maximum of 54 (severe depression).
Time Frame: 8 weeks
Population: QEEG data were collected, analyzed and reported as part of a larger trial. The analysis of QEEG data per protocol was only possible using the proprietary algorithm developed by a company; acquisition of that company precludes analysis for this study alone. Larger study reported in: Iosifescu DV et al. Eur Neuropsychopharmacol. 2009;19:772-7.
Arm/Group | Open-label Selective Serotonin Reuptake Inhibitor (SSRI)
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Time Frame: 8 weeks
Arm/Group | Open-label SSRI
Serious Adverse Events (participants affected / at risk) | 0/47
Other Adverse Events (participants affected / at risk) | 5/47
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Open-label SSRI (N=47)
weight gain (Metabolism and nutrition disorders) | 1 (1)
lack of appetite (Metabolism and nutrition disorders) | 1 (1)
increase in tremors (Musculoskeletal and connective tissue disorders) | 1 (1)
nausea (Gastrointestinal disorders) | 1 (1)
hypomania (Psychiatric disorders) | 1 (1)

LIMITATIONS AND CAVEATS:
For the secondary outcome measure, the data were analyzed and reported as part of a larger trial; however, because the analysis could only be done using a proprietary algorithm, the subset for this study could not be independently analyzed.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No